CLINICAL TRIAL: NCT01410422
Title: Exhaled Breath Analysis in Patients With COPD and Bronchiectasis
Brief Title: Metabolomic Analysis of Exhaled Breath Condensates in Patients With COPD and Bronchiectasis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Ping-Hung Kuo, MD., National Taiwan University Hospital
Other Study IDs: 201103010RC
Record Dates: First submitted 2011-08-04; First posted 2011-08-05 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2011-05

CONDITIONS: COPD; Bronchiectasis
Keywords: COPD; Bronchiectasis; Metabolomics
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchiectasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Breath condensate, blood, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- COPD: COPD
- Bronchiectasis: Bronchiectasis

SUMMARY:
Metabolomics is a large-scale approach to monitoring the compounds involved in cellular processes. It may reflect changes in biological function. Collection of exhaled breath is a newly developed, noninvasive method that may allow clinicians and researchers to assess biochemical profiles in the airway. This study is conducted for the metabolomic analysis of the exhaled gas in patients with Chronic Obstructive Pulmonary Disease (COPD) and bronchiectasis.

DETAILED DESCRIPTION:
Metabolomics is a large-scale approach to monitoring as many as possible of the compounds involved in cellular processes in a single assay to derive metabolic profiles. Compared with genomics or proteomics, metabolomics reflects changes in phenotype and therefore function. Collection of exhaled breath condensate (EBC) is a newly developed, noninvasive method that may allow clinicians and researchers to assess biochemical profiles in the alveolar lining fluid. The aims of this study are: (1)Collecting and metabolomic profiling of the EBCs from patients with COPD/bronchiectasis; (2) Comparing the profiles of these patients obtained during stable and acute exacerbation periods; (3) Comparing the profiles of these patients with and without Pseudomonas colonization/infection; (4) Correlation of EBC metabolomic profiles with clinical phenotypes, severity and outcomes of these patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with COPD or bronchiectasis

Exclusion Criteria:

* not willing to sign ICF

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COPD and bronchiectasis
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2011-05; Study Completion 2014-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ping-Hung Kuo, M.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan